CLINICAL TRIAL: NCT03815058
Title: A Phase II, Open-Label, Multicenter, Randomized Study of the Efficacy and Safety of RO7198457 in Combination With Pembrolizumab Versus Pembrolizumab in Patients With Previously Untreated Advanced Melanoma
Brief Title: A Study to Evaluate the Efficacy and Safety of Autogene Cevumeran (RO7198457) in Combination With Pembrolizumab Versus Pembrolizumab Alone in Participants With Previously Untreated Advanced Melanoma.
Acronym: IMCODE001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO40558; 2018-001773-24 (EudraCT Number); 2023-507389-15-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2019-01-07; First posted 2019-01-24 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Advanced Melanoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety Run-in Period: Autogene Cevumeran + Pembrolizumab (Experimental): Participants will receive at least one cycle of 200 mg pembrolizumab monotherapy by intravenous (IV) infusion followed by 200 mg pembrolizumab IV infusion every 3 weeks (Q3W) plus a recommended dose of autogene cevumeran.
  Interventions: Biological: Autogene cevumeran; Drug: Pembrolizumab
- Randomized Period: Arm A: Pembrolizumab (Active Comparator): Participants will receive 200 mg pembrolizumab administered by IV infusion Q3W. Participants in Arm A have the option to cross over to combination treatment with autogene cevumeran plus pembrolizumab (Arm B) after confirmed disease progression.
  Interventions: Drug: Pembrolizumab
- Randomized Period: Arm B: Autogene Cevumeran + Pembrolizumab (Experimental): Participants will receive at least one cycle of 200 mg pembrolizumab monotherapy by IV infusion followed by 200 mg pembrolizumab IV infusion Q3W plus a recommended dose of autogene cevumeran.
  Interventions: Biological: Autogene cevumeran; Drug: Pembrolizumab

INTERVENTIONS:
Biological: Autogene cevumeran — Participants will receive a recommended dose of autogene cevumeran administered by IV infusion at protocol-defined intervals.
  Other Names: RO7198457
  Arms: Randomized Period: Arm B: Autogene Cevumeran + Pembrolizumab; Safety Run-in Period: Autogene Cevumeran + Pembrolizumab
Drug: Pembrolizumab — Participants will receive 200 mg pembrolizumab administered by IV infusion Q3W.
  Other Names: Keytruda

SUMMARY:
This study will evaluate the efficacy, safety, pharmacokinetics, and patient-reported outcomes (PROs) of autogene cevumeran (RO7198457) plus pembrolizumab compared with pembrolizumab alone in patients with previously untreated advanced melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic (recurrent or de novo Stage IV) or unresectable locally advanced (Stage IIIC or IIID) cutaneous, acral, or mucosal melanoma;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
* Life expectancy >/= 12 weeks;
* Adequate hematologic and end-organ function;
* Naive to prior systemic anti-cancer therapy for advanced melanoma with some exceptions;
* Tumor specimen availability;
* Measurable disease per RECIST v1.1.

Exclusion criteria:

* Ocular/uveal melanoma;
* Any anti-cancer therapy with the exceptions as specified in the protocol;
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases;
* Previous splenectomy;
* History of autoimmune disease;
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation;
* Positive test for Human Immunodeficiency Virus (HIV) infection;
* Active hepatitis B or C or tuberculosis;
* Significant cardiovascular disease;
* Known clinically significant liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (41):
- United States (17):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - UCSF Comprehensive Cancer Ctr, San Francisco, California
  - University of Colorado, Denver, Colorado
  - Cancer Specialists, Jacksonville, Florida
  - Moffitt McKinley Outpatient Center, Tampa, Florida
  - Atlanta Cancer Care, Alpharetta, Georgia
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital., Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Case Western Research University, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
  - Intermountain Surgical Oncology, Murray, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (5):
  - Liverpool Hospital, Liverpool, New South Wales
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - St. John of God - Subiaco Hospital, Subiaco, Western Australia
- Belgium (2):
  - Antwerp University Hospital, Edegem
  - ZAS Sint Augustinus Wilrijk, Wilrijk
- Germany (9):
  - Elbe Kliniken Stade-Buxtehude GmbH, Buxtehude
  - Universitätsklinikum Koeln, Cologne
  - Universitatsklinikum Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Uni Schleswig-Holstein, Lübeck
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz KöR, Hautklinik und Poliklinik, Mainz
  - Med. Fakultat Mannheim der Universitat Heidelberg, Mannheim
  - Fachklinik Hornheide, Münster
  - Universitätshautk. Tübingen, Tübingen
- Spain (7):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Instituto Oncológico Dr. Rosell, Barcelona
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- Barts and The London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 131 participants with previously untreated advanced melanoma took part in the study at 40 investigative sites across the United States, Germany, Australia, Spain, Belgium, and the United Kingdom from 21 December 2018 to 21 January 2025. The study consists of an initial safety run-in stage followed by a randomized stage (Arm A & Arm B). Participants in Arm A had an option to crossover to Arm B after confirmed disease progression (PD), if crossover eligibility criteria were met.
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive either pembrolizumab (Arm A) or pembrolizumab + RO7198457 (Arm B). 1 participant in Arm A did not receive any study treatment and was excluded from safety analysis. 4 participants in Arm B discontinued study treatment after receiving pembrolizumab but prior to receiving RO7198457 & were therefore considered in Arm A for safety analysis.
Groups:
- Safety Run-in: Participants received pembrolizumab monotherapy, 200 milligrams (mg) as an intravenous (IV) infusion for at least 1 cycle, followed by pembrolizumab, 200 mg, IV infusion, every 3 weeks (Q3W) thereafter, along with RO7198457. Participants received RO7198457, 25 micrograms (µg), as an IV infusion, 4 doses every week (QW) and 4 doses Q3W as induction dosing and then maintenance dosing every 8 cycles until the occurrence of unacceptable toxicity or PD or death, whichever occurred first (1 cycle = 21 days).
- Arm A: Pembrolizumab: Participants received pembrolizumab, 200 mg, as an IV infusion, Q3W until the occurrence of unacceptable toxicity or PD or death, whichever occurred first.
- Arm B: Pembrolizumab + RO7198457: Participants received pembrolizumab, 200 mg, as an IV infusion for at least 1 cycle (1 cycle = 21 days), followed by pembrolizumab, 200 mg, Q3W along with RO7198457. Participants received RO7198457, 25 µg, as an IV infusion, 4 doses QW and 4 doses Q3W as induction dosing and then maintenance dosing, every 8 cycles until the occurrence of unacceptable toxicity or PD or death, whichever occurred first (1 cycle = 21 days).
- Crossover: Pembrolizumab + RO7198457: Participants in Arm A with confirmed PD were given the option to crossover & receive RO7198457 in combination with pembrolizumab, 200 mg, as an IV infusion, Q3W. Participants received RO7198457, 25 µg, as an IV infusion, 4 doses QW and 4 doses Q3W as induction dosing and then maintenance dosing, every 8 cycles until the occurrence of unacceptable toxicity or PD or death, whichever occurred first (1 cycle = 21 days).
Period: Safety Run-in Stage
Arm/Group | Safety Run-in | Arm A: Pembrolizumab | Arm B: Pembrolizumab + RO7198457 | Crossover: Pembrolizumab + RO7198457
Started | 6 | 0 | 0 | 0
Safety-evaluable (SE) Population (SE population included all participants who received at least 1 dose of study treatment.) | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0
Not completed — Study Ended by Sponsor | 4 | 0 | 0 | 0
Period: Randomized Stage
Arm/Group | Safety Run-in | Arm A: Pembrolizumab | Arm B: Pembrolizumab + RO7198457 | Crossover: Pembrolizumab + RO7198457
Started | 0 | 41 | 84 | 0
SE Population (SE population included all participants who received at least 1 dose of study treatment.) | 0 | 44 | 80 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 41 | 84 | 0
Not completed — Death | 0 | 13 | 29 | 0
Not completed — Lost to Follow-up | 0 | 2 | 4 | 0
Not completed — Study Ended by Sponsor | 0 | 14 | 42 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 9 | 0
Not completed — Discontinued due to PD to Receive Cross-over Treatment | 0 | 10 | 0 | 0
Period: Cross-over Treatment
Arm/Group | Safety Run-in | Arm A: Pembrolizumab | Arm B: Pembrolizumab + RO7198457 | Crossover: Pembrolizumab + RO7198457
Started | 0 | 0 | 0 | 10
SE Population (SE population included all participants who received at least 1 dose of study treatment.) | 0 | 0 | 0 | 10
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 10
Not completed — Death | 0 | 0 | 0 | 2
Not completed — Study Ended by Sponsor | 0 | 0 | 0 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Safety Run-in: Participants received pembrolizumab monotherapy, 200 mg as an IV infusion for at least 1 cycle, followed by pembrolizumab, 200 mg, IV infusion, Q3W thereafter, along with RO7198457. Participants received RO7198457, 25 µg, as an IV infusion, 4 doses QW and 4 doses Q3W as induction dosing and then maintenance dosing every 8 cycles until the occurrence of unacceptable toxicity or PD or death, whichever occurred first (1 cycle = 21 days).
- Total: Total of all reporting groups
Arm/Group | Safety Run-in | Arm A: Pembrolizumab | Arm B: Pembrolizumab + RO7198457 | Total
Number analyzed (Participants) | 6 | 41 | 84 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (11.0) | 62.4 (14.4) | 63.6 (14.2) | 63.2 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 11 | 27 | 39
  Male | 5 | 30 | 57 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 39 | 69 | 114
  Unknown or Not Reported | 0 | 1 | 14 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 6 | 38 | 80 | 124
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v.1.1) After Randomization
Description: PFS was defined as the time from randomization to the first documented PD as determined by the investigator according to RECIST v1.1 or death from any cause, whichever occurred first. PD was defined as at least a 20% increase in the sum of diameters (SOD) of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). Kaplan-Meier (KM) method was used to estimate median PFS.
Time Frame: From randomization to PD or death (up to approximately 60 months)
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pembrolizumab | Arm B: Pembrolizumab + RO7198457
Number analyzed (Participants) | 41 | 84
months | 7.9 [2.8 to 22.7] | 8.3 [6.9 to 26.9]
Statistical Analysis 1: Comparison: Arm A: Pembrolizumab vs Arm B: Pembrolizumab + RO7198457; Test type: Superiority; p = 0.3284, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.49 to 1.27]

2. Secondary Outcome: Objective Response Rate (ORR) According to RECIST V.1.1 After Randomization
Description: ORR was defined as the percentage of participants with a complete response (CR) or a partial response (PR) on two consecutive occasions ≥ 4 weeks apart, as determined by the investigator according to RECIST v1.1. CR was defined as the disappearance of all target lesions or any pathological lymph nodes must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. Percentages have been rounded off to the nearest whole number.
Time Frame: Up to approximately 60 months
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Pembrolizumab | Arm B: Pembrolizumab + RO7198457
Number analyzed (Participants) | 41 | 84
percentage of participants | 48.8 [32.26 to 65.30] | 41.7 [30.53 to 52.80]

3. Secondary Outcome: Overall Survival (OS) After Randomization
Description: OS was defined as the time from randomization to death from any cause. KM method was used to estimate the median OS.
Time Frame: From randomization to death (up to approximately 63 months)
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pembrolizumab | Arm B: Pembrolizumab + RO7198457
Number analyzed (Participants) | 41 | 84
months | NA [19.6 to NA] — The median and upper limit of the 95% confidence interval (CI) were not estimable due to an insufficient number of participants with events. | 62.2 [41.8 to NA] — The upper limit of the 95% CI was not estimable due to an insufficient number of participants with events.

4. Secondary Outcome: Duration of Response (DOR) According to RECIST V.1.1 After Randomization
Description: DOR was defined as the time from the first occurrence of a documented objective response (OR) to PD or death from any cause, whichever occurred first, as determined by the investigator according to RECIST v1.1. CR was defined as the disappearance of all target lesions or any pathological lymph nodes must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. DOR was estimated using the KM methodology.
Time Frame: Up to approximately 60 months
Population: ITT population included all randomized participants. Overall number analyzed is the number of participants with an OR (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Pembrolizumab | Arm B: Pembrolizumab + RO7198457
Number analyzed (Participants) | 20 | 35
months | NA [19.8 to NA] — The median and upper limit of the 95% CI were not estimable due to an insufficient number of participants with events. | NA [36.1 to NA] — The median and upper limit of the 95% CI were not estimable due to an insufficient number of participants with events.

5. Secondary Outcome: Change From Baseline in Global Health Status (GHS)/Health-related Quality of Life (HRQoL) Score Assessed by European Organisation for Research and Treatment of Cancer 30-Item Quality of Life Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 consists of 30 questions that assess participant functioning (physical, emotional, role, cognitive, and social), symptom scales (fatigue, nausea and vomiting, pain), GHS/QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Change in HRQoL was assessed using participant responses to questions regarding GHS (Question 29: GHS; "How would you rate your overall health during the past week?") and QoL (Question 30: QoL; "How would you rate your overall quality of life during the past week?") and were scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores were standardized. Scores range from 0-100. A higher score indicates a better QoL.
Time Frame: Baseline, Day 1 of Cycles 1 to 34, time of first PD, time to last dose, treatment discontinuation and study drug completion (up to approximately 29 months) (1 cycle = 21 days)
Population: ITT population included all randomized participants. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Pembrolizumab | Arm B: Pembrolizumab + RO7198457
Number analyzed (Participants) | 39 | 83
score on a scale
  Baseline | 64.74 (24.67) | 73.39 (21.56)
  Change at Cycle 1 Day 1: number analyzed (Participants) | 0 | 83
  Change at Cycle 1 Day 1 |  | 0.00 (0.00)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 36 | 79
  Change at Cycle 2 Day 1 | -1.85 (17.72) | -1.37 (14.40)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 32 | 77
  Change at Cycle 3 Day 1 | 2.60 (16.73) | 0.54 (16.69)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 29 | 72
  Change at Cycle 4 Day 1 | 3.74 (16.45) | -3.70 (19.48)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 26 | 68
  Change at Cycle 5 Day 1 | 3.53 (19.32) | -1.84 (15.56)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 22 | 65
  Change at Cycle 6 Day 1 | 0.00 (20.57) | -6.03 (22.51)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 22 | 58
  Change at Cycle 7 Day 1 | 2.27 (15.04) | -1.01 (15.85)
  Change at Cycle 8 Day 1: number analyzed (Participants) | 20 | 54
  Change at Cycle 8 Day 1 | 0.83 (10.08) | 0.15 (18.35)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 20 | 49
  Change at Cycle 9 Day 1 | -2.92 (12.76) | -1.19 (15.77)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 19 | 47
  Change at Cycle 10 Day 1 | 4.39 (14.26) | -3.72 (15.43)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 16 | 47
  Change at Cycle 11 Day 1 | 0.52 (16.52) | 1.06 (14.29)
  Change at Cycle 12 Day 1: number analyzed (Participants) | 16 | 43
  Change at Cycle 12 Day 1 | 1.56 (13.34) | -4.07 (14.82)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 15 | 43
  Change at Cycle 13 Day 1 | 1.11 (24.57) | 0.00 (13.61)
  Change at Cycle 14 Day 1: number analyzed (Participants) | 14 | 41
  Change at Cycle 14 Day 1 | 2.98 (12.49) | -2.03 (13.54)
  Change at Cycle 15 Day 1: number analyzed (Participants) | 15 | 38
  Change at Cycle 15 Day 1 | 0.56 (13.16) | -3.07 (16.37)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 13 | 34
  Change at Cycle 16 Day 1 | 0.64 (16.12) | -1.72 (15.04)
  Change at Cycle 17 Day 1: number analyzed (Participants) | 12 | 32
  Change at Cycle 17 Day 1 | 4.86 (15.27) | -2.60 (15.62)
  Change at Cycle 18 Day 1: number analyzed (Participants) | 10 | 31
  Change at Cycle 18 Day 1 | 5.00 (18.51) | -4.57 (17.72)
  Change at Cycle 19 Day 1: number analyzed (Participants) | 10 | 31
  Change at Cycle 19 Day 1 | 0.00 (19.64) | -1.61 (14.18)
  Change at Cycle 20 Day 1: number analyzed (Participants) | 9 | 30
  Change at Cycle 20 Day 1 | 5.56 (11.79) | -1.67 (14.42)
  Change at Cycle 21 Day 1: number analyzed (Participants) | 9 | 27
  Change at Cycle 21 Day 1 | 9.26 (12.80) | -0.31 (15.41)
  Change at Cycle 22 Day 1: number analyzed (Participants) | 8 | 28
  Change at Cycle 22 Day 1 | 11.46 (12.55) | -1.79 (17.18)
  Change at Cycle 23 Day 1: number analyzed (Participants) | 9 | 28
  Change at Cycle 23 Day 1 | 8.33 (9.32) | -2.68 (17.43)
  Change at Cycle 24 Day 1: number analyzed (Participants) | 9 | 28
  Change at Cycle 24 Day 1 | 2.78 (13.82) | -3.87 (22.28)
  Change at Cycle 25 Day 1: number analyzed (Participants) | 9 | 26
  Change at Cycle 25 Day 1 | 1.85 (18.53) | -4.81 (18.59)
  Change at Cycle 26 Day 1: number analyzed (Participants) | 8 | 27
  Change at Cycle 26 Day 1 | 5.21 (14.04) | -3.40 (14.85)
  Change at Cycle 27 Day 1: number analyzed (Participants) | 8 | 27
  Change at Cycle 27 Day 1 | 0.00 (8.91) | -2.47 (15.64)
  Change at Cycle 28 Day 1: number analyzed (Participants) | 7 | 25
  Change at Cycle 28 Day 1 | -4.76 (20.89) | -2.67 (17.47)
  Change at Cycle 29 Day 1: number analyzed (Participants) | 8 | 27
  Change at Cycle 29 Day 1 | 2.08 (14.60) | -2.47 (15.98)
  Change at Cycle 30 Day 1: number analyzed (Participants) | 8 | 26
  Change at Cycle 30 Day 1 | -1.04 (5.34) | -7.69 (17.47)
  Change at Cycle 31 Day 1: number analyzed (Participants) | 8 | 25
  Change at Cycle 31 Day 1 | 3.13 (14.73) | -3.67 (18.65)
  Change at Cycle 32 Day 1: number analyzed (Participants) | 8 | 26
  Change at Cycle 32 Day 1 | 7.29 (14.39) | -3.21 (18.72)
  Change at Cycle 33 Day 1: number analyzed (Participants) | 8 | 26
  Change at Cycle 33 Day 1 | 5.21 (13.32) | -4.81 (18.59)
  Change at Cycle 34 Day 1: number analyzed (Participants) | 8 | 25
  Change at Cycle 34 Day 1 | 7.29 (13.68) | -5.00 (18.16)
  Change at Time of First PD: number analyzed (Participants) | 17 | 40
  Change at Time of First PD | -1.47 (26.06) | -4.17 (19.43)
  Change at Time of Last Dose: number analyzed (Participants) | 31 | 81
  Change at Time of Last Dose | -5.65 (25.40) | -7.30 (23.55)
  Change at Treatment Discontinuation: number analyzed (Participants) | 22 | 64
  Change at Treatment Discontinuation | -2.27 (26.75) | -11.07 (18.43)
  Change at Study Drug Completion: number analyzed (Participants) | 0 | 0

6. Secondary Outcome: ORR According to RECIST V.1.1 After Crossover
Description: ORR was defined as the percentage of participants with a CR or PR on two consecutive occasions ≥ 4 weeks apart, as determined by the investigator according to RECIST v1.1. CR was defined as disappearance of all target lesions or any pathological lymph nodes must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR.
Time Frame: Up to 54.7 months
Population: Crossover ITT population included all randomized participants who entered crossover period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Crossover: Pembrolizumab + RO7198457
Number analyzed (Participants) | 10
percentage of participants | 40.0 [4.64 to 75.36]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.
Time Frame: Baseline up to 90 days after the final dose of study drug (Safety run-in and randomized stage: up to 32 months; Cross-over stage: up to 24 months)
Population: SE population included all participants who received at least 1 dose of study treatment. 1 participant in Arm A didn't receive any study treatment & was excluded from safety. 4 participants in Arm B discontinued study treatment after receiving pembrolizumab but prior to receiving RO7198457 & were therefore considered in Arm A for safety analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Safety Run-in: Participants received pembrolizumab monotherapy, 200 mg, as an IV infusion for at least 1 cycle, followed by pembrolizumab, 200 mg as an IV infusion, Q3W thereafter, along with RO7198457. Participants received RO7198457, 25 µg, IV infusion, 4 doses QW and 4 doses Q3W as induction dosing and then maintenance dosing every 8 cycles until the occurrence of unacceptable toxicity or PD or death, whichever occurred first (1 cycle = 21 days).
Arm/Group | Safety Run-in | Arm A: Pembrolizumab | Arm B: Pembrolizumab + RO7198457 | Crossover: Pembrolizumab + RO7198457
Number analyzed (Participants) | 6 | 44 | 80 | 10
Participants | 6 | 43 | 79 | 10

ADVERSE EVENTS:
Time Frame: Baseline up to 90 days after the final dose of study drug (Safety run-in and randomized stage: up to 32 months; Cross-over stage: up to 24 months); All-cause Mortality: up to approximately 63 months
Description: Safety-evaluable population included all participants who received at least 1 dose of study treatment. 1 participant in Arm A did not receive any study treatment & was excluded from safety analysis. 4 participants in Arm B discontinued study treatment after receiving pembrolizumab but prior to receiving RO7198457 & were therefore considered in Arm A for safety analysis.
Arm/Group | Safety Run-in | Arm A: Pembrolizumab | Arm B: Pembrolizumab + RO7198457 | Crossover: Pembrolizumab + RO7198457
All-Cause Mortality (participants affected / at risk) | 2/6 | 14/44 | 30/80 | 3/10
Serious Adverse Events (participants affected / at risk) | 3/6 | 16/44 | 25/80 | 4/10
Other Adverse Events (participants affected / at risk) | 6/6 | 40/44 | 78/80 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-in (N=6) | Arm A: Pembrolizumab (N=44) | Arm B: Pembrolizumab + RO7198457 (N=80) | Crossover: Pembrolizumab + RO7198457 (N=10)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Human bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5) | 3 (3) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated encephalitis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-in (N=6) | Arm A: Pembrolizumab (N=44) | Arm B: Pembrolizumab + RO7198457 (N=80) | Crossover: Pembrolizumab + RO7198457 (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 12 (18) | 1 (2)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (6) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 8 (9) | 3 (3)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 5 (7) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 8 (10) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 2 (2) | 9 (9) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Vision blurred (Eye disorders) | 0 (0) | 5 (5) | 4 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 6 (6) | 8 (8) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Anal rash (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 7 (8) | 10 (11) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 10 (14) | 23 (36) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 8 (8) | 7 (7) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 5 (5) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4) | 11 (14) | 22 (33) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (4) | 1 (1) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (6) | 4 (6) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (5) | 11 (13) | 1 (1)
Asthenia (General disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (4) | 4 (4) | 1 (2)
Chills (General disorders) | 2 (2) | 1 (1) | 3 (4) | 1 (1)
Fatigue (General disorders) | 5 (5) | 13 (16) | 36 (48) | 5 (6)
Influenza like illness (General disorders) | 3 (15) | 4 (5) | 14 (54) | 1 (5)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 7 (8) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (2) | 7 (8) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 3 (16) | 0 (0) | 2 (2) | 1 (5)
Drug hypersensitivity (Immune system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 13 (16) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 8 (9) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 13 (17) | 1 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 7 (13) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 62 (251) | 5 (17)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access site erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (4) | 8 (9) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 3 (3) | 10 (14) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (5) | 7 (7) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (3) | 5 (13) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 3 (3) | 11 (20) | 1 (3)
Weight decreased (Investigations) | 1 (1) | 3 (3) | 6 (6) | 0 (0)
Weight increased (Investigations) | 0 (0) | 2 (3) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 10 (14) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (9) | 0 (0) | 2 (12)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (4) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 3 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (2) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (9) | 20 (25) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (8) | 7 (10) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (9) | 12 (12) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 7 (7) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 7 (7) | 1 (1)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 3 (3) | 7 (12) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 3 (3) | 15 (22) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 5 (5) | 5 (5) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Renal cyst haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (9) | 13 (13) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 10 (11) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 10 (13) | 11 (12) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (8) | 16 (18) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (5) | 5 (7) | 8 (10) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 9 (9) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 5 (6) | 9 (13) | 4 (6)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 1 (2) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT03815058/Prot_SAP_000.pdf